CLINICAL TRIAL: NCT00323128
Title: Validation of Serum Creatinine Dosage and Renal Clearance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Arjan Van Der Tol, University Hospital Ghent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006/037
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Calculation of inuline clearance — Calculation of inuline clearance.
Procedure: Measuring serum creatinine — Measuring serum creatinine.

SUMMARY:
This study has an open study design. The GFR will be measured using the renal clearance of inulin (Inutest) in volunteers with different stage of renal disease or without renal disease. A blood sample will be obtained for measuring serum creatinine in different laboratories.

DETAILED DESCRIPTION:
In this study we will investigate the correlation between the GFR as measured by inulin clearance (golden standard) and the estimated GFR as measured by laboratories which used different serum creatinine assays in patients without renal disease and in patients with different stage of kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight as defined by a Body Mass Index of 18 to 30 kg/m2.
* Subject is competent and willing to sign informed consent form after being given all the detailed information about the study. Informed consent form signed voluntarily.
* The subjects must be in stable clinical condition, with stable serum creatinin at least for 6 months.
* Persons with different stage of chronic renal disease and without kidney disease (living donors) who need an evaluation of the GFR or Admitted volunteers who easily obtain urine samples.

Exclusion Criteria:

* Transplant patients
* Medication that will influence the serumcreatinine.
* Morbid obesity
* Pregnant, lactating females or females with childbearing potential without adequate contraception (use of oral contraceptives, IUD or condoms with spermicide).
* History of allergy or hypersensitivity to inulin
* Donation of blood in the 60 days preceding the first visit.
* Liver disease, heart failure, nephrotic syndrome.
* Patients in critically ill conditions.
* Malnutrition
* Postrenal kidney failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration ratio | At time T0
Serum creatinine | At time T0

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Van Holder, MD, PhD, Principal Investigator — University Hospital, Ghent; Arjan Van der Tol, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be